CLINICAL TRIAL: NCT00913601
Title: Treatment of Idiopathic Faecal Incontinence With Sacral Nerve Stimulation - Improved Function With Implantation and Stimulation of Permanent Electrodes Bilaterally - a Double-blinded Randomized Cross-over Trial
Brief Title: Treatment of Faecal Incontinence With Sacral Nerve Stimulation - Improved Function With Stimulation Bilaterally?
Acronym: SNS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Prematurely stopped, as no beneficial effect was evident for bilateral stimulation after interim analysis of the first 20 patients.
Sponsor: University of Aarhus (Other)
Collaborators: MEDTRONIC DANMARK A/S Arne Jacobsens Alle 17 DK-2300 København S Danmark (Unknown)
Responsible Party: Principal Investigator, Jakob Jakobsen, M.D., University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Fecal Incontinence
Keywords: Idiopathic Fecal Incontinence; Fecal Incontinence; Sacral Nerve Stimulation; Sacral Nerve Neuromodulation
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dextra (Experimental): Unilateral sacral nerve stimulation dextra for 4 weeks
  Interventions: Device: Medtronic INTERSIM II - 3058
- Sinistra (Experimental): Unilateral sacral nerve stimulation sinistra 4 weeks
  Interventions: Device: Medtronic INTERSIM II - 3058
- Bilateral (Experimental): Bilateral sacral nerve stimulation 4 weeks
  Interventions: Device: Medtronic INTERSIM II - 3058

INTERVENTIONS:
Device: Medtronic INTERSIM II - 3058 — Medtronic INTERSIM II - 3058 Impuls Generator
  Other Names: Impuls Generator

SUMMARY:
Faecal incontinence is a devastating condition causing psychological stress, affecting daily living and influences quality of life. Faecal incontinence affects 2,2 to 5 % of the adult population. The magnitude of the problem is probably underestimated, because most patients don't discuss this affliction with their general practitioner. A new treatment, sacral nerve stimulation (SNS), has over the last decade given hope to these patients. The treatment is divided in two; first a test operation (PNE-test) has to reveal if the patient will benefit from treatment with permanent sacral nerve stimulation. Second if the patient benefit from the PNE-test, they proceed to final implant. 75-80% of the patients with idiopathic fecal incontinence benefit from the PNE-test, 70% of those get satisfactory functional results and the remaining 30% get suboptimal improvement in continence after permanent unilateral sacral nerve stimulation. The aim of this project is to investigate if bilateral sacral nerve stimulation can produce better fecal continence results than standard unilateral stimulation, through a double blind, randomized crossover study.

DETAILED DESCRIPTION:
Sacral nerve stimulation is a very good and effective treatment for faecal incontinence The method was introduced to patients with voiding disorders in 1981. In 1995 sacral nerve stimulation was used for three patients with faecal incontinence, two were afterwards fully continent. The method has over the last decade been used increasingly in Europe. The method is now used routinely in the treatment of faecal incontinence in Europe.

Recent studies have shown that the effect of sacral nerve stimulation is due to a neuromodulation in the central nervous system, whereas direct stimulation of efferent nerves to anal sphincter and the pelvic floor has less significance.

The sacral nerve stimulation is performed in two steps, first a test stimulation, if positive the patients proceed to permanent implant.

Test stimulation (PNE-test) is performed over a 3 week period. If this test stimulation produces a decrease in incontinence episodes of more than 50 per cent, a permanent electrode and neurostimulator are implanted. The test period has a success rate of approximately 75-80% in patients with idiopathic fecal incontinence or incontinence after anal surgery. These 75-80% will normal be candidates to unilateral implantation of permanent electrode and neurostimulator.

All permanently implanted has less incontinence symptoms after the treatment. Satisfactory continence results after permanent implantation are seen in 70% of the patients, the remaining 30% only obtain a suboptimal efficacy. It is unclear whether these patients could have a more optimal function if they were stimulate on more than one sacral nerve simultaneously.

Hypothesis: Is it possible to improve the functional result in faecal incontinent patients treated with routine unilateral sacral nerve stimulation by stimulating the sacral nerves bilaterally.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Diagnosed with idiopathic faecal incontinence and planned sacral nerve stimulation
* Age> 40 years normal sigmoid/colonoscopic prior to operation

Exclusion Criteria:

* Pregnant or breastfeeding
* Patients who are not deemed able to follow the planned testing program, including mental illness or mentally unstable patients
* Medication with known effects on gastrointestinal motility, thyroid disease, diabetes, coeliaki, neurological disorders.
* Irritable Bowel Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-05; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of faecal incontinence episodes per week. | 1, 2, and 3 months after enrolment to the project

SECONDARY OUTCOMES:
Days with faecal soiling. | 1, 2, and 3 months after enrolment to the project
Days with faecal urgency. | 1, 2, and 3 months after enrolment to the project
Wexner incontinence score. | 1, 2, and 3 months after enrolment to the project
Anal physiological changes during SNS bilateral versus unilateral. | 1, 2, and 3 months after enrolment to the project
Quality of life assessment (Rockwood - Fecal incontinence quality of life) | 1, 2, and 3 months after enrolment to the project

CONTACTS AND LOCATIONS:
Overall Officials: Jakob K Jakobsen, MD, Principal Investigator — Anal Physiology Laboratory, Surgical Research Section 900, Aarhus University Hospital, Denmark
Locations (1):
- Anal Physiology Laboratory, Surgical Research Section 900, Aarhus University Hospital, Aarhus, Aarhus C, Denmark

REFERENCES:
- [Background] Matzel KE, Stadelmaier U, Hohenfellner M, Gall FP. Electrical stimulation of sacral spinal nerves for treatment of faecal incontinence. Lancet. 1995 Oct 28;346(8983):1124-7. doi: 10.1016/s0140-6736(95)91799-3. PMID 7475602
- [Background] Vaizey CJ, Kamm MA, Turner IC, Nicholls RJ, Woloszko J. Effects of short term sacral nerve stimulation on anal and rectal function in patients with anal incontinence. Gut. 1999 Mar;44(3):407-12. doi: 10.1136/gut.44.3.407. PMID 10026329
- [Background] Rasmussen OO, Christiansen J. [Sacral nerve stimulation in fecal incontinence]. Ugeskr Laeger. 2002 Aug 12;164(33):3866-8. Danish. PMID 12216156
- [Background] Jarrett ME, Mowatt G, Glazener CM, Fraser C, Nicholls RJ, Grant AM, Kamm MA. Systematic review of sacral nerve stimulation for faecal incontinence and constipation. Br J Surg. 2004 Dec;91(12):1559-69. doi: 10.1002/bjs.4796. PMID 15455360
- [Background] Michelsen HB, Buntzen S, Krogh K, Laurberg S. Rectal volume tolerability and anal pressures in patients with fecal incontinence treated with sacral nerve stimulation. Dis Colon Rectum. 2006 Jul;49(7):1039-44. doi: 10.1007/s10350-006-0548-8. PMID 16721520